CLINICAL TRIAL: NCT07291557
Title: PSMA-PET Directed Radiation Therapy in High and Very High-Risk Prostate Cancer
Brief Title: PSMA-PET Directed Radiation Therapy for High-Risk Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0031
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Radiotherapy; PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate Only Radiation Therapy (PORT) (Active Comparator): Radiation therapy: prostate and surrounding tissues
  Interventions: Radiation: Prostate Only Radiation Therapy (PORT)
- Prostate + Whole Pelvis Radiation Therapy (P-WPRT) (Experimental): Radiation therapy: prostate and surrounding tissues + whole pelvis radiation therapy
  Interventions: Radiation: Prostate + Whole Pelvis Radiation Therapy (P-WPRT)

INTERVENTIONS:
Radiation: Prostate Only Radiation Therapy (PORT) — 6800cGy in 25 daily fractions to the prostate and surrounding tissues
  Arms: Prostate Only Radiation Therapy (PORT)
Radiation: Prostate + Whole Pelvis Radiation Therapy (P-WPRT) — 6800cGy to the prostate and surrounding tissues + 5000cGy to the whole pelvis in 25 daily fractions.
  Arms: Prostate + Whole Pelvis Radiation Therapy (P-WPRT)

SUMMARY:
In this study, prostate cancer patients whose cancer has not spread to the lymph nodes will receive radiation therapy targeted to the prostate and nearby tissues with or without whole pelvis radiation therapy. PSMA imaging will be used to visualize prostate cancer prior to starting the trial.

DETAILED DESCRIPTION:
The current treatment of high risk and very high risk localized prostate cancer is by radiation therapy (RT) and hormone therapy (ADT). RT uses radiation to kill the cancer cells while hormone therapy lowers the levels of male hormones like testosterone, which the cancer needs to grow. Radiation is targeted to the prostate and nearby tissues, which may or may not include whole pelvis radiation therapy (WPRT). The benefit of whole pelvis radiation therapy is not well understood. Therefore, clinical research is needed to assess the benefits/risks of whole pelvis radiation therapy in prostate cancer treatment. In addition to traditional cancer imaging methods like CT, MRI, and bone scan, new techniques like PSMA imaging are now available to examine prostate cancer. The PSMA scan involves a small amount of radioactive tracer (18F-PSMA-1007) being injected into the vein, which marks the prostate cancer cells for better visualization of the cancer location and spread. Because of its higher accuracy, results of PSMA scans can change how doctors plan cancer treatment, like where they aim radiation and how much they use.

In this study, prostate cancer patients whose cancer has not spread to the lymph nodes will receive radiation therapy. PSMA imaging will be used to visualize prostate cancer prior to starting the trial.

There will be two treatment groups (1) Prostate Only Radiation Therapy (PORT), and Prostate + Whole Pelvis Radiation Therapy (P-WPRT), and all participants will receive hormone therapy as part of standard of care. In addition to comparing the biochemical failure free survival (BFFS) between the two treatment groups, the study will also compare distant metastases free survival (DMFS), toxicity, patient reported outcomes and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

PSMA-N0M0 patients who have a documented history of High Risk localized adenocarcinoma of the prostate are eligible to participate if they meet the following eligibility criteria:

1. Participants capable of giving written informed consent.
2. Male.
3. Age ≥18 years.
4. ECOG ≤2.
5. Patient has histologically proven adenocarcinoma of prostate gland with an assigned Gleason score and Gleason Grade Group.
6. ≥NCCN High-Risk localized disease as per standard imaging investigations including pelvic imaging (CT, MRI) and 99Tc bone scan. High Risk prostate cancer defined as any of the following: cT3-T4 disease OR PSA ≥20 ng/ml OR Gleason grade group 4 or 5.
7. No documentation of regional nodal (N1) or metastatic (M1) prostate cancer on standard imaging (CT, MRI, or 99Tc bone scan).
8. In the opinion of the treating oncologist, patient is fit to undergo radical external beam radiotherapy to the prostate.
9. Patient commits to androgen suppression treatment as per standard of care. 10. Patient is willing to complete symptom and patient reported outcome questionnaires.

11. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 6 months after the last dose of radiation therapy. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.

Male patients should agree to not donate sperm during the study and for 6 months after completion of radiation therapy.

Exclusion Criteria:

1. Inability to complete the investigational imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.).
2. Any additional medical condition, serious inter-current illness or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study performance, interpretation, or compliance with radiation
3. Patients who have initiated therapy (ADT, systemic therapy, or radiation) for their prostate cancer prior to PSMA-PET imaging.
4. History of inflammatory bowel disease, anal stenosis, colorectal surgery, or repeated endoscopic examinations/interventions related to anorectal diseases.
5. History of prostatectomy or previous pelvic radiotherapy.
6. Previous malignancy within the last five years, except BCC or SCC skin or a malignancy treated curatively with no evidence of disease for ≥5 years.
7. Bilateral hip prostheses will be ineligible for study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2031-05 (Estimated); Study Completion 2036-05 (Estimated)

PRIMARY OUTCOMES:
5-year Biochemical Failure Free Survival (BFFS) | Number of events as measured from the date of randomization to 5-years.
  As measured from the date of randomization to the first recorded date of biochemical failure as defined by serum PSA exceeding nadir PSA +2 ng/mL.

SECONDARY OUTCOMES:
Distant metastases-free survival (DMFS) | As measured from the date of randomization until the development of first distant metastasis outside the pelvic nodal regions or date of death from any cause, whichever came first; assessed up to 10 years (end of extended follow-up)
  Calculated from the time of randomization until the development of first distant metastasis outside the pelvic nodal regions. Patients will be censored at either the date of last follow-up or date of death.
Acute and late toxicity as per CTCAE 5.0 | Acute toxicity will be measured up to the 90 days post-radiation, and late toxicity will be monitored over the course of the study follow-up, up to 5 years post-radiation.
  Patient toxicity will be documented as per the domains of the CTCAE v5.0.
Overall survival | As measured form the time of randomization to date of death from any cause, assessed up to 10 years (end of extended follow-up)
  As measured form the time of randomization to the time of death from any cause.
Patient reported outcomes: IPSS | Outcomes will be measured from the completion of radiation up to 90 days post-radiation, and over the course of the study follow-up, up to 5 years post-radiation.
  International Prostate Symptom Score (IPSS) is a standardized questionnaire used worldwide to assess the severity of urinary symptoms. It consists of 7 questions, each scored from 0 (no symptoms) to 5 (most severe symptoms). The total score is the sum of all responses, giving a range from 0 to 35
Patient reported outcomes: EQ-5D | Outcomes will be measured from the completion of radiation up to 90 days post-radiation, and over the course of the study follow-up, up to 5 years post-radiation.
  The 5-item EQ-5D index score will be transformed into a utility score between 0, "Worst health state," and 1, "Best health state." The index score or the cost-utility equation can be used in the quality adjusted survival analysis. For this study, the plan is to report the multidimensional utilities for comparative purposes.
Patient reported outcomes: EPIC-26 | Outcomes will be measured from the completion of radiation up to 90 days post-radiation, and over the course of the study follow-up, up to 5 years post-radiation.
  Expanded Prostate Cancer Index Composite - Short Form (EPIC-26) uses a 0-100 scale per domain, where 0 means worst function and 100 means best function. EPIC-26 overall score will be reported, as well as intra-individual change from baseline. Score changes will also be stratified by clinically minimally important differences of 5 for bowel and hormonal, 7 for urinary, and 10 for sexual domain

OTHER OUTCOMES:
10-year Biochemical Failure Free Survival (BFFS) | Retrospective chart reviews will occur during long term follow-up (years 5 to 10, inclusive).
  Patient charts will be reviewed retrospectively after patients have completed clinical trial follow-up for clinical history up to 10 years postradiation. BFFS will be calculated from the time of randomization to the date to PSA relapse
10-year Disease Free Survival (DFS) | Retrospective chart reviews will occur during long term follow-up (years 5 to 10, inclusive).
  Patient charts will be reviewed retrospectively after patients have completed clinical trial follow-up for clinical history up to 10 years postradiation. DFS is calculated from the time of randomization to the first biochemical or clinicoradiological recurrence of disease at any site, or death due to any cause, whichever occurs earlier
10-year Distant Metastases-Free Survival (DMFS) | Retrospective chart reviews will occur during long term follow-up (years 5 to 10, inclusive).
  Patient charts will be reviewed retrospectively after patients have completed clinical trial follow-up for clinical history up to 10 years postradiation. DMFS will be calculated from the time of randomization until the development of first distant metastasis outside the pelvic nodal regions.
Assessment of fatigue over the course of therapy | Outcomes will be measured from the completion of radiation up to 90 days post-radiation, and over the course of the study follow-up, up to 5 years post-radiation.
  Patient level of fatigue will be assessed as a patient reported outcome using the validated Brief Fatigue Inventory (BFI) which will be completed at each of the AE and quality of life assessments. BFI uses a 0-10 scale per item, with 0 meaning no fatigue and 10 meaning the worst fatigue. Longitudinal scores for each patient will be correlated with therapy received and radiation dosimetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No